CLINICAL TRIAL: NCT02385097
Title: A Prospective, Randomised, Non-inferiority Study of Chloroprocaine 2% and the Active Control Ropivacaine 0.75% (AstraZeneca) in Ultrasound-guided Axillary Nerve Block for Short-duration Distal Upper Limb Surgery
Brief Title: Chloroprocaine 2% vs Ropivacaine 0.75% in Ultrasound-guided Axillary Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Collaborators: Cross S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CHL.2/01-2014/M
Record Dates: First submitted 2015-02-20; First posted 2015-03-11 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Axillary Nerve Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroprocaine HCl 2% (20 mg/mL) (Experimental): Chloroprocaine 2 % Solution for injection, single administration by axillary nerve route 20 mL
  Interventions: Drug: Chloroprocaine HCl 2%
- Ropivacaine 0.75% (7.5 mg/mL) (Active Comparator): Ropivacaine 0.75% Solution for injection, single administration by axillary nerve route 20 mL
  Interventions: Drug: Ropivacaine 0.75%

INTERVENTIONS:
Drug: Chloroprocaine HCl 2% — Single Administration (20mL) by Axillary Nerve Route
  Other Names: Ampres
  Arms: Chloroprocaine HCl 2% (20 mg/mL)
Drug: Ropivacaine 0.75% — Single Administration (20mL) by Axillary Nerve Route
  Other Names: Naropin
  Arms: Ropivacaine 0.75% (7.5 mg/mL)

SUMMARY:
The Study evaluate the non-inferiority of Test product (Chloroprocaine 2%) versus Reference product (Ropivacaine 0.75%) in terms of proportion of subjects with a successful block for distal upper limb surgeries Successful block: anaesthesia adequate for the surgery without any supplementation in the first 45 min.

DETAILED DESCRIPTION:
This Study evaluate the non-inferiority of Test product (Chloroprocaine 2%) versus Reference product (Ropivacaine 0.75%) in terms of proportion of subjects with a successful block for distal upper limb surgeries, without any supplementation in the first 45 min (see definitions below), calculated from the time of readiness for surgery (complete sensory block). Successful block: anaesthesia adequate for the surgery (complete sensory block), without any supplementation in the first 45 min (even if surgery lasts for > 45 min), calculated from the time of readiness for surgery (complete sensory block). Supplementation: i.v. premedication or general anaesthesia or pre- or intra-operative systemic analgesia or additional local anaesthetic infiltration

ELIGIBILITY:
Inclusion Criteria:

1. Sex and surgery: male and female patients scheduled for short duration (< 60 min) distal upper limb surgery under axillary nerve block anaesthesia
2. Age: ≥ 18 years old
3. Body Mass Index (BMI): 18 - 32 kg/m2 inclusive
4. ASA physical status: I-III
5. Informed consent: signed written informed consent before inclusion in the study
6. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study

Exclusion Criteria:

1. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study. Contraindications to peripheral nerve block anaesthesia. History of neuromuscular diseases to the upper extremities
2. Axillary status: Axillary local infections, surgical scarring and pathological lymph node enlargement
3. ASA physical status: IV-V
4. Further anaesthesia: Patients anticipated to be requiring further anaesthesia (general or local anaesthesia)
5. Chronic pain syndromes: Patients with chronic pain syndromes (taking opioids, antidepressants, anticonvulsant agents)
6. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations ingredients; ascertained or presumptive hypersensitivity to the amide and ester-type anaesthetics
7. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; ascertained psychiatric diseases, sepsis, blood coagulation disorders, insulin dependent diabetes mellitus, terminal kidney failure
8. Medications: Medication known to interfere with the extent of regional blocks (see chloroprocaine and ropivacaine SmPCs) for 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
9. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study, calculated from the first day of the month following the last visit of the previous study
10. Drug, alcohol: history of drug or alcohol abuse
11. Pregnancy: missing or positive pregnancy test at screening, pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, Prof, Principal Investigator — Department of General Anesthesia and Intensive Care Medicine, Spitalgasse 23, 1090 Vienna, Austria; Claudio Camponovo, MD, Principal Investigator — Department of Anaesthesiology,Clinica Ars Medica,Via Cantonale, CH-6929 Gravesano, Switzerland; Andrea Saporito, MD, Principal Investigator — Department of Anaesthesiology, Ospedale Regionale di Bellinzona, CH-6500 Bellinzona, Switzerland
Locations (1):
- Claudio Camponovo, Gravesano, Lugano, Switzerland

REFERENCES:
- [Derived] Sulyok I, Camponovo C, Zotti O, Haslik W, Kostenberger M, Likar R, Leuratti C, Donati E, Kimberger O. A randomised, non-inferiority study of chloroprocaine 2% and ropivacaine 0.75% in ultrasound-guided axillary block. Sci Rep. 2021 May 11;11(1):10035. doi: 10.1038/s41598-021-89483-y. PMID 33976374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2015 to May 2017 in Medical clinic and Hospital
Period: Overall Study
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Started | 106 | 105
Completed | 106 | 105
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 211 patients were enrolled in the study. 106 of the enrolled patients were randomised to the Test treatment group and 105 patients to the Reference treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL) | Total
Number analyzed (Participants) | 106 | 105 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (15.4) | 52.6 (18.7) | 54 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 60 | 131
  Male | 35 | 45 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 104 | 101 | 205
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 62 | 62 | 124
  Switzerland | 44 | 43 | 87
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.58 (3.83) | 25.61 (3.55) | 25.60 (3.69)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Block for Distal Upper Limb Surgeries
Description: Percentage of patients with a successful block for distal upper limb surgeries, without any supplementation in the first 45 min, calculated from the time of readiness for surgery (complete sensory block).
Time Frame: 45 min from the time of readiness of surgery
Population: 211 patients were enrolled in the study. 106 of the enrolled patients were randomised to the Test treatment group and 105 patients to the Reference treatment group. Two subjects, one in the Test and one in the Reference treatment group discontinued the study before treatment (withdrawal by subject). In the Test treatment group, 105 patients were treated and completed the study. In the Reference treatment group, 104 patients were treated, 103 of them completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
Participants | 96 | 97

2. Secondary Outcome: Time to Onset of Sensory Block (Corresponding to Readiness for Surgery)
Description: Time period from completion of the final perineural injection (time 0 h) to achievement of sensory block in the 4 nerve territories
Time Frame: Up to 1 h after last perineural injection
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
minutes | 10 [10 to 15] | 15 [10 to 15]

3. Secondary Outcome: Time to Onset of Motor Block
Description: Time period from completion of the final perineural injection (time 0 h) to achievement of motor block
Time Frame: Up to 1 h after last perineural injection
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
minutes | 10 [5 to 10] | 10 [5 to 10]

4. Secondary Outcome: Time to Regression of Sensory Block
Description: Will be deemed to have occurred when cold sensation and sensitive perception have returned (if assessable) in any nerve territory
Time Frame: Up to 12 hrs after surgery
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
minutes | 68 [64 to 75] | 451 [413 to 480]

5. Secondary Outcome: Time to Regression of Motor Block
Description: Will be deemed to have occurred when motor score is ≥ 3 (Modified Bromage scale) in any nerve territory (Modified Bromage scale: 0-No movement in relevant muscle group,1-Flicker of movement in relevant muscle group,2-Ability to move relevant muscle group against gravity but inability to move against resistance,3-Reduced power but ability to move muscle group against resistance,4-Full power in relevant muscle group)
Time Frame: Up to 12 hrs after surgery
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
minutes | 65 [60 to 69] | 415 [388 to 460]

6. Secondary Outcome: Partecipants Received Rescue Anaesthesia or Rescue Analgesia
Description: partecipants received rescue anaesthesia or rescue analgesia from completion of the final perineural injection (time 0 hour) to administration of first rescue anaesthesia or analgesia (supplementation)
Time Frame: 45 min from the time of readiness of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
Participants | 9 | 7

7. Secondary Outcome: Number of Subjects Who Received Post-operative Analgesia
Description: Number of subjects who received the first post-operative analgesia
Time Frame: From surgery day to 24 hrs post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
Participants | 49 | 46

8. Secondary Outcome: Time to Eligibility for Home Discharge
Description: Time from completion of the final perineural injection (time 0 h) to the time when the criteria for discharge are met, even if, according to the hospital procedures, the patient is discharged from the hospital at a later time
Time Frame: from surgery day to 24h post surgery
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
minutes | 161 [155 to 170] | 355.5 [260 to 450]

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of Participants with Treatment-emergent Adverse Events (TEAEs) occurring or worsening after the first dose of IMP
Time Frame: from surgery day to day 6 +/- 1 after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
Participants | 58 | 76

10. Secondary Outcome: Neurological Symptoms
Description: Number of patients with Neurological Symptoms (e.g. paraesthesia, motor function problems and pain at the injection site)
Time Frame: from surgery day to day 6 +/- 1 after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
Participants
  burning : discharge | 8 | 1
  burning : day 7 | 6 | 4
  tingling : discharge | 8 | 25
  tingling : day 7 | 5 | 6
  Pins and needles sensation : discharge | 1 | 5
  Pins and needles sensation : day 7 | 2 | 0
  Pricking : discharge | 8 | 5
  Pricking : day 7 | 0 | 0
  aching : discharge | 10 | 6
  aching : day 7 | 4 | 3
  numbness : discharge | 2 | 27
  numbness : day 7 | 2 | 3
  hypoesthesia : discharge | 5 | 14
  hypoesthesia : day 7 | 5 | 5
  Pain surgery site : discharge | 0 | 1
  Pain surgery site : day 7 | 0 | 0
  diffuse hair loss : discharge | 0 | 0
  diffuse hair loss : day 7 | 0 | 1
  headache : discharge | 0 | 0
  headache : day 7 | 2 | 0
  itching : discharge | 0 | 0
  itching : day 7 | 0 | 1

11. Secondary Outcome: Heart Rate
Description: The following normal ranges Heart Rate parameters will be used:
  50-90 beats/min
Time Frame: from surgery day to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: beats/minutes
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
beats/minutes
  screening | 73 (12) | 73.6 (12.3)
  baseline | 72.5 (10.8) | 71.6 (12.5)
  discharge | 71.5 (11.5) | 73 (12.3)

12. Secondary Outcome: Blood Pressure
Description: The following normal ranges Systolic and Diastolic Blood Pressure parameters will be used:
  Systolic Blood Pressure: 100-139 mmHg Diastolic Blood Pressure: 50-89 mmHg
Time Frame: from surgery day to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
mmHg
  Systolic Blood Pressure at screening | 137 (20.5) | 136.2 (18.2)
  Systolic Blood Pressure at baseline | 136.6 (18.9) | 138 (19.1)
  Systolic Blood Pressure at discharge | 130.5 (17.8) | 130.1 (17.3)
  Diastolic Blood Pressure at screening | 80.8 (11.4) | 80.5 (9.8)
  Diastolic Blood Pressure at baseline | 78.2 (10.7) | 80.1 (10.4)
  Diastolic Blood Pressure at discharge | 74.4 (11.1) | 75.4 (9.8)

13. Secondary Outcome: SpO2
Description: The following normal ranges SpO2 parameters will be used:
  Peripheral Oxygen Saturation: ≥ 95%
Time Frame: from surgery day to 24 hrs post surgery
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
percentage of SpO2
  baseline | 97.05 (1.51) | 97.36 (1.69)
  discharge | 97.47 (1.52) | 97.61 (1.33)

14. Secondary Outcome: Number of Participants With Normal Electrocardiogram (ECG) Parameters
Description: Number of Participants with Normal Electrocardiogram (ECG) Parameters. The following normal ranges ECG parameters will be used:
  Heart Rate: 50-90 beats/min PR Interval: 100-220 msec QRS Duration: ≤ 120 msec QT Interval: ≤ 500 msec
Time Frame: from surgery day to 24 hrs post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
Number analyzed (Participants) | 105 | 104
Participants | 105 | 104

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Chloroprocaine HCl 2% (20 mg/mL) | Ropivacaine 0.75% (7.5 mg/mL)
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/105
Other Adverse Events (participants affected / at risk) | 58/106 | 76/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroprocaine HCl 2% (20 mg/mL) (N=106) | Ropivacaine 0.75% (7.5 mg/mL) (N=105)
Procedural pain (Injury, poisoning and procedural complications) | 48 (50) | 41 (43)
Hypoaestesia (Nervous system disorders) | 9 (10) | 38 (44)
Paraestesia (Nervous system disorders) | 17 (22) | 28 (40)
burning sensation (Nervous system disorders) | 11 (11) | 5 (5)
headache (Nervous system disorders) | 3 (3) | 1 (1)
sensorimotor disorder (Nervous system disorders) | 0 (0) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12) | 5 (5)
injection site pain (General disorders) | 6 (6) | 5 (5)
nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT02385097/Prot_SAP_000.pdf